CLINICAL TRIAL: NCT00004729
Title: Efficacy of the Ketogenic Diet -- a Blinded Study
Brief Title: Ketogenic Diet for Child Epilepsy and Seizure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS035980 (NIH)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Epilepsy; Seizures; Lennox-Gastaut Syndrome
Keywords: child; children; epilepsy; seizure; ketogenic; diet; Lennox-Gastaut Syndrome; LGS
MeSH Terms: conditions — Epilepsy; Seizures; Lennox Gastaut Syndrome | interventions — Diet, Ketogenic

INTERVENTIONS:
Behavioral: Ketogenic diet

SUMMARY:
Twenty to thirty percent of children with epilepsy continue to suffer from seizures, even when treated with currently available anticonvulsant medications. Children with Lennox-Gastaut Syndrome (LGS) are particularly handicapped by atonic-myoclonic seizures. Preliminary data suggest that even when other medications have failed, these seizures may respond rapidly and dramatically to a high-fat-low-carbohydrate ketogenic diet. The purpose of the study is to assess if the classic ketogenic diet is efficacious in reducing seizure frequency, medication toxicity, and improves quality of life.

DETAILED DESCRIPTION:
The ketogenic diet (KD) is a form of therapy for seizures that involves a brief period of fasting followed by a very carefully controlled high fat-low protein and carbohydrate diet. Studies suggest it is useful in children whose seizures could not be controlled by any of the medicines available. This study is designed to test, in a carefully controlled fashion, how well the diet works in children with "drop" seizures. Children who experience 15 or more drop seizures each day, despite having used at least two medications, may be eligible to participate. This study requires children to undergo periods of fasting and to maintain a carefully controlled diet. Parents of participating children monitor their children's diets and keep daily meal and seizure diaries.

ELIGIBILITY:
Inclusion Criteria:

* >15 myoclonic or atonic seizures a day
* EEG with Lennox-Gastaut pattern

Exclusion Criteria:

* <15 atonic or myoclonic seizures a day
* on >3 medications
* previously on diet and/or evidence of metabolic disorder

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1997-07

CONTACTS AND LOCATIONS:
Overall Officials: John M. Freeman, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States